CLINICAL TRIAL: NCT06236594
Title: Application of Multimodal Endoscopic Functional Imaging Technology in the Diagnosis of Common Gastrointestinal Diseases
Acronym: Endo-mmfi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: multimodal endoscopic imaging
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Gastrointestinal Disease
Keywords: endoscopic laser speckle imaging; multispectral blood oxygen imaging; gastrointestinal lesions; early diagnosis; gastrointestinal tumors
MeSH Terms: conditions — Gastrointestinal Diseases; Disease; Digestive System Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After the acquisition of endoscopic images, endoscopic pathological biopsy is routinely performed for patients who consider the presence of mucosal lesions. Endoscopic mucosal resection (EMR) or submucosal dissection (ESD) is performed for inpatients in the Department of Gastroenterology according to clinical needs, and postoperatively the specimens will be sent to the Department of Pathology for further pathological analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We plan the study to explore the application of endoscopic laser speckle imaging and multispectral blood oxygen imaging to observe gastrointestinal lesions, as well as the differences in the morphology, density and functional status of mucosal surfaces and deep blood vessels of different gastrointestinal lesions, also to explore the role of endoscopic multimodal functional imaging in common gastrointestinal diseases, especially in the early diagnosis of gastrointestinal tumors.

DETAILED DESCRIPTION:
The current focus of electronic endoscopy is on the morphology and fine structure of the mucosal surface, and there is no effective observation method for the deep structure of the mucosa and the function of blood oxygen binding. However, the multilayer morphology and functions of mucosal vessels under different conditions of digestive tract lesions should be different. Therefore, we propose a method of endoscopic multimodal functional imaging to the conventional endoscopic examinations observing the mucosa of the digestive tract, which is based on the existing electronic endoscope, laser speckle contrast imaging and multispectral blood oxygen imaging technology. Laser irradiation was given to obtain the information of coherent light on the mucosal surface and deep scattering of coherent light to obtain multi-level vascular distribution information, and multispectral irradiation imaging was carried out to obtain the oxygenation situation of the mucosa. Finally, we may find the differences of images of deep blood vessels among common gastrointestinal diseases, which could help us to make early diagnosis of gastrointestinal tumors noninvasively.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old, gender is not limited
2. Diagnosed or suspected of one of the following common gastrointestinal mucosal diseases: Chronic non-atrophic gastritis, chronic atrophic gastritis, gastric polyps, early gastric cancer, advanced gastric cancer, colon polyps, colon melanosis, inflammatory bowel disease, early colon cancer, advanced colon cancer
3. Sign the informed consent form -

Exclusion Criteria:

1. Combined with cardiovascular and cerebrovascular diseases, or severe impairment of liver, kidney and hematopoietic system;
2. mentally ill;
3. the presence of bleeding disorders;
4. Platelet count<50×10^9/L;
5. Inability to tolerate or cooperate with endoscopy;
6. Patients with serious complications, such as severe infection, gastrointestinal bleeding, obstruction, perforation, etc.;
7. Pregnant or lactating women.
8. Refuse to sign the informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Image quality rate | one year
  The main evaluation index (image quality rate) is based on FAS(Full Analysis Set) and PPS(Per Protocol Set), for statistical description. Image quality rate Calculation formula: image excellent rate = number of cases with excellent or good image quality evaluation ÷ number of subjects undergoing multimodal endoscopy × 100%.

SECONDARY OUTCOMES:
Diagnosis accuracy according to image | one year
  (1) Endoscopy examinations combined with laser speckle imaging and Doppler blood oxygen imaging can realize multi-level vascular observation and photographing of the mucosa, and the imaging analyzer will analyzes and synthesizes the two-dimensional map of laser speckle and blood oxygen imaging of the mucosa. Endoscopist will make diagnosis according to the image they get. (2) After endoscopic biopsy or endoscopic mucosal resection (EMR), endoscopic submucosal resection (ESD) obtaining tissue specimens, the pathology was observed by conventional HE staining or immunohistochemistry. (3) The results of comparison are divided into conformity, partial conformity and non-conformity.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China